CLINICAL TRIAL: NCT04054024
Title: A Placebo-Controlled, Double-Blind, Randomized, Proof-of-Concept Study to Evaluate the Efficacy and Tolerability of Erenumab in Patients With Trigeminal Neuralgia
Brief Title: Efficacy and Tolerability of Erenumab in Patients With Trigeminal Neuralgia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Stine Maarbjerg, MD, Principal investigator, Danish Headache Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-19011013
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — erenumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Placebo is saline
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active drug (Active Comparator)
  Interventions: Drug: Erenumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Erenumab — 140 mg Erenumab
  Arms: Active drug
Drug: Placebos — Saline
  Arms: Placebo

SUMMARY:
A placebo-controlled, double-blind, randomized proof-of-concept study to evaluate the efficacy and tolerability of the CGRP receptor antibody erenumab in treating pain experienced by subjects with TN.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of primary TN (idiopathic or classical) according to criteria of The Interna-tional Classification of Headache Disorders 3rd edition (1).
* Age between 18 and 85 years.
* Subjects must have a minimum mean of three TN related pain paroxysms per day with a mean ADP of 4 to 10, inclusive, on the 11-point NRS (0= no pain; 10= maximum pain imaginable) during the 7-day screening phase to enter the baseline phase.
* Subjects must have a minimum mean of three TN related pain paroxysms per day with a mean ADP of 4 to 10, inclusive, on the 11-point NRS (0= no pain; 10= maximum pain imaginable) during the 4-week baseline phase to enter the treatment phase (to be randomized).
* Fertile women must use safe contraceptives and present with a negative u-HCG at visit 1. Safe contraceptives are defined as intra-uterine devices, contraceptive pills or implants and surgical sterilization.

Exclusion Criteria:

* Significant cardiovascular and cerebrovascular disease such as ischemic heart disease, previous myocardial infarction or previous stroke or transient ischemic attack, major CVD interventions.
* Language difficulties.
* Poor compliance, i.e. unlikely to be able to complete all protocol required study visits or procedures, and/or to comply with all required study procedures to the best of the sub-ject's and investigator's knowledge.
* Severe psychiatric disease.
* Anamnestic or clinical symptoms of any kind that are deemed relevant for study partici-pation by the physician who examines the patient.
* Taking any TN-medication, where the prescribed daily dose has changed within 2 weeks prior to the baseline period (refer to section 6.4 for the list of these medications).
* Pregnant or breastfeeding, or is a female expecting to conceive during the study, includ-ing through 4 weeks after treatment.
* Female subject of childbearing potential who is unwilling to use an acceptable method of effective contraception during the study. Acceptable methods of effective birth control include not having intercourse (true abstinence, when this is in line with the preferred and usual lifestyle of the subject), hormonal birth control methods (pills, shots/injections, implants, or patches), intrauterine devices, surgical contraceptive methods (vasectomy with medical assessment of the surgical success of this procedure or bilateral tubal ligation), or two barrier methods (each partner must use one barrier method) with spermicide - males must use a condom with spermicide; females must choose either a diaphragm with spermicide, OR cervical cap with spermicide, OR contraceptive sponge with spermicide. Female subjects not of childbearing potential are defined as any female who: is post-menopausal by history, defined as:

Age ≥ 55 years with cessation of menses for 12 or more months, OR Age < 55 years but no spontaneous menses for at least 2 years, OR Age < 55 years and spontaneous menses within the past 1 year, but currently amenorrheic (eg, spontaneous or secondary to hysterectomy), AND with postmenopausal gonadotro-pin levels (luteinizing hormone and follicle-stimulating hormone levels > 40 IU/L) or postmenopausal estradiol levels (< 5 ng/dL) or according to the definition of "postmeno-pausal range" for the laboratory involved. OR o Underwent bilateral oophorectomy OR o Underwent hysterectomy OR o Underwent bilateral salpingectomy.

* Known sensitivity to any component of erenumab.
* Member of investigational site staff or relative of the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects classified as responders at the end of the evaluation period. | 4 weeks after randomization
  A subject who meets the following criterion will be classified as a responder:
  Has a reduction of ≥ 30% in mean average daily pain intensity score (mean ADP) assessed using the 11-point numerical rating scale (NRS) during the evaluation period (week 1-4) compared with baseline (weeks -4 to -1). Patients that are protocol violators, e.g., patients having to increase current medications or undergoes surgery in the evaluation period as well as pa-tients who drop out due to worsening of symptoms or side effects will be recorded as non-responders.

SECONDARY OUTCOMES:
Secondary outcome measures | 4 weeks after randomization
  1. proportion of subjects reaching ≥50% reduction in mean ADP (average daily pain) during the evaluation period (week 1-4) compared with baseline (week -4 to -1).
  2. proportion of subjects reaching ≥75% reduction in mean ADP during the evaluation period (week 1-4) compared with baseline (week -4 to -1).
  3. subjects with a response in number of paroxysms at evaluation period.
  4. proportion of subjects with a Patient Global Impression of Change (PGIC) scale response at evaluation period.
  Due to word limitations not all secondary outcome measures were explaned in detail and/or registered.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Bendtsen, MD, Dr Med Sci, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Department of Neurology, Rigshospitalet - Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided